CLINICAL TRIAL: NCT00006252
Title: Minimal Ablation and Cellular Immune Therapy of Chronic Lymphocytic Leukemia, Prolymphocytic Leukemia, Low-Grade Non-Hodgkin's Lymphoma, and Mantle Cell Lymphoma With Allogeneic Donor Stem Cells
Brief Title: Fludarabine and Cyclophosphamide Followed by Peripheral Stem Cell Transplant in Treating Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer and Leukemia Group B (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Alliance for Clinical Trials in Oncology (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-109901; U10CA031946 (NIH); CALGB-109901; CDR0000068185 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; prolymphocytic leukemia; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — fludarabine phosphate; Cyclophosphamide; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogeneic Stem Cell Tx (Experimental): minimal ablation and cellular immune therapy with allogeneic donor stem cell therapy
  Interventions: Drug: fludarabine phosphate; Drug: Cyclophosphamide; Biological: PBSC; Drug: G-CSF; Biological: Donor lymphocytes

INTERVENTIONS:
Drug: fludarabine phosphate — 30 mg/sq m/day IV infusion for 5 days (Days -7 thru -3)
Drug: Cyclophosphamide — 1 g/sq m/day IV infusion x 3 days (Days -5 thru -3)
Biological: PBSC — 2-8,000,000/kg CD34+ cells via infusion on Day 0
Drug: G-CSF — 5 ug/kg/day subQ injection until ANC > 1000/uL for 3 days beginning Day 5
Biological: Donor lymphocytes — 10,000,000 CD3+ cells/kg via infusion

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as fludarabine and cyclophosphamide, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well fludarabine and cyclophosphamide followed by peripheral stem cell transplant works in treating patients with leukemia or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of fludarabine and cyclophosphamide followed by allogeneic peripheral blood stem cell transplantation, in terms of 6-month treatment-related mortality, in patients with chronic lymphocytic leukemia, prolymphocytic leukemia, low-grade non-Hodgkin's lymphoma, or mantle cell lymphoma.
* Determine the 6-month and 12-month probabilities of response in patients treated with this regimen.
* Determine the time to disease progression in patients responding to this regimen.
* Determine the percentage of donor chimerism achieved in patients treated with this regimen.
* Determine the risk of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the overall survival and disease-free survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive fludarabine IV over 30 minutes on days -7 to -3 and cyclophosphamide IV over 1 to 2 hours on days -5 to -3. Patients undergo allogeneic peripheral blood stem cell transplantation on days 0-1. Patients then receive filgrastim (G-CSF) subcutaneously daily beginning on day 5 and continuing until blood counts recover.

Patients with no signs of active graft-versus host disease and stable or progressive disease receive donor lymphocytes IV over 2 hours beginning after day 120. Patients may receive a total of 3 infusions at least 8 weeks apart if disease remains stable or progressive.

Patients are followed every 3 months for 2 years and then every 6 months for 5 years.

PROJECTED ACCRUAL: A maximum of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses:

  * Chronic lymphocytic leukemia

    * Absolute lymphocytosis greater than 5,000/mm^3
    * Morphologically mature lymphocytes with less than 55% prolymphocytes
    * Lymphocyte phenotypic expression of CD19 and CD5
    * Failed at least 1 prior regimen

      * Progressive lymphocytosis with more than 50% increase in peripheral lymphocytosis or a progressive lymph node or spleen enlargement (at least 25% enlargement or the appearance of new lymph nodes) that persists for at least 4 weeks despite concurrent or prior drug treatment OR
    * At least 1 of the following high-risk factors and not in first complete remission

= 17p deletion = 11q deletion

* Unmutated VH gene status
* p53 mutations

  * Prolymphocytic leukemia (PLL)

    * Absolute lymphocytosis greater than 5,000/mm^3
    * Morphologically mature lymphocytes with more than 55% prolymphocytes
  * Low-grade non-Hodgkin's lymphoma

    * Small lymphocytic lymphoma
    * Follicular center lymphoma (grade I or II)
    * Diffuse (predominately small cell type)
    * Marginal zone, B-cell lymphoma
    * No transformed lymphoma
    * Failure of at least 1 prior regimen OR
    * At least 3 of the following risk factors:
* Over 60 years of age
* Performance status greater than 1
* LDH greater than normal
* More than 1 site of extranodal disease
* Disease stage III or IV

  * Mantle cell lymphoma

    * Any stage
    * Ineligible for protocol CALGB-59908
    * At least 1 prior treatment regimen
    * At least 1 of the following:
* Immunophenotypic expression of CD5 and CD19 and absence of CD23
* Cytogenetic analysis with presence of t(11;14)
* Overexpression of cyclin D1
* Rearrangement of BCL1 gene

  * Responsive or stable disease to most recent prior therapy

    * Prior therapy for PLL not required
  * Must have HLA identical sibling (6/6) donor by serologic typing (A, B, DR)

    * No syngeneic donors
    * No age restriction NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* Under 70

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 500/mm^3*
* Platelet count at least 50,000/mm^3* NOTE: *Unless attributable to disease

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)*
* AST no greater than 3 times ULN* NOTE: *Unless attributable to disease

Renal:

* Creatinine clearance at least 40 mL/min, unless attributable to disease

Cardiovascular:

* LVEF at least 30% by MUGA

Pulmonary:

* DLCO greater than 40%
* No symptomatic pulmonary disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled diabetes mellitus
* No active serious infection
* No known hypersensitivity to E. coli-derived products

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior autologous transplantation

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* At least 4 weeks since prior surgery

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2001-02; Primary Completion 2007-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality within the first 6 months post-transplant | 6 months post chemo initiation

SECONDARY OUTCOMES:
Response | 6 months & 12 months
Percentage of patients achieving complete donor chimerism or mixed donor chimerism | 90 days post transplant
Survival | 5 years post study entry
  Disease free and overall survival will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Shea, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (19):
- United States (19):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Cancer Institute of New Jersey at the Cooper University Hospital - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Mount Sinai Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Shea T, Johnson J, Westervelt P, Farag S, McCarty J, Bashey A, Isola L, Baxter-Lowe LA, Kelly M, Owzar K, Linker C; Cancer and Leukemia Group B. Reduced-intensity allogeneic transplantation provides high event-free and overall survival in patients with advanced indolent B cell malignancies: CALGB 109901. Biol Blood Marrow Transplant. 2011 Sep;17(9):1395-403. doi: 10.1016/j.bbmt.2011.01.016. Epub 2011 Feb 3. PMID 21296675